CLINICAL TRIAL: NCT00018655
Title: Integrated Intervention for Substance Abusers With Depressive Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MHBS-041-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Substance-Related Disorders; Depressive Disorder
Keywords: Mood Disorders; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders; Depressive Disorder; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Twelve Step Facilitation
  Interventions: Behavioral: Twelve Step Facilitation
- Arm 2 (Experimental): Integrated Cognitive Behavioral Treatment
  Interventions: Behavioral: Integrated Cognitive Behavioral Treatment

INTERVENTIONS:
Behavioral: Twelve Step Facilitation — Twelve Step Facilitation Therapy involves focusing on topics from 12-Step programs which support sobriety goals and personal growth.
  Arms: Arm 1
Behavioral: Integrated Cognitive Behavioral Treatment — Integrated Cognitive Behavioral Treatment involves focusing on thoughts, activities, and interactions with people related to depressive symptoms and/or substance use.
  Arms: Arm 2

SUMMARY:
This study is a randomized clinical trial comparing outcomes of Integrated Cognitive Behavioral Treatment plus standard medications for veterans with both substance use disorders, depressive disorders versus the most commonly administered form of therapy for substance use disorders and depression, Twelve Step Facilitation (AA/NA model) group treatment plus medications.

DETAILED DESCRIPTION:
This study is a randomized clinical trial comparing outcomes of Integrated Cognitive Behavioral Treatment plus standard medications for veterans with both substance use disorders, depressive disorders versus the most commonly administered form of therapy for substance use disorders and depression, Twelve Step Facilitation (AA/NA model) group treatment plus medications. Follow-up assessments were conducted at quarterly intervals for one year following treatment.

ELIGIBILITY:
Inclusion Criteria:

Veterans age 18 and older with alcohol, cannabinol, and/or stimulant dependence and independent mood disorders will be included.

Exclusion Criteria:

Psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2000-04; Primary Completion 2009-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale, Timeline Follow-back (substance measure) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tate, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Brown SA, Glasner-Edwards SV, Tate SR, McQuaid JR, Chalekian J, Granholm E. Integrated cognitive behavioral therapy versus twelve-step facilitation therapy for substance-dependent adults with depressive disorders. J Psychoactive Drugs. 2006 Dec;38(4):449-60. doi: 10.1080/02791072.2006.10400584. PMID 17373561
- [Result] Drapkin ML, Tate SR, McQuaid JR, Brown SA. Does initial treatment focus influence outcomes for depressed substance abusers? J Subst Abuse Treat. 2008 Oct;35(3):343-50. doi: 10.1016/j.jsat.2007.12.005. Epub 2008 Mar 4. PMID 18295436
- [Result] Glasner-Edwards S, Tate SR, McQuaid JR, Cummins K, Granholm E, Brown SA. Mechanisms of action in integrated cognitive-behavioral treatment versus twelve-step facilitation for substance-dependent adults with comorbid major depression. J Stud Alcohol Drugs. 2007 Sep;68(5):663-72. doi: 10.15288/jsad.2007.68.663. PMID 17690799
- [Result] Lydecker KP, Tate SR, Cummins KM, McQuaid J, Granholm E, Brown SA. Clinical outcomes of an integrated treatment for depression and substance use disorders. Psychol Addict Behav. 2010 Sep;24(3):453-65. doi: 10.1037/a0019943. PMID 20853931
- [Result] Granholm E, Tate SR, Link PC, Lydecker KP, Cummins KM, McQuaid J, Shriver C, Brown SA. Neuropsychological functioning and outcomes of treatment for co-occurring depression and substance use disorders. Am J Drug Alcohol Abuse. 2011 Jul;37(4):240-9. doi: 10.3109/00952990.2011.570829. Epub 2011 Apr 26. PMID 21517712
- [Result] Tate SR, Mrnak-Meyer J, Shriver CL, Atkinson JH, Robinson SK, Brown SA. Predictors of treatment retention for substance-dependent adults with co-occurring depression. Am J Addict. 2011 Jul-Aug;20(4):357-65. doi: 10.1111/j.1521-0391.2011.00137.x. Epub 2011 May 31. PMID 21679267
- [Result] Worley MJ, Trim RS, Roesch SC, Mrnak-Meyer J, Tate SR, Brown SA. Comorbid depression and substance use disorder: longitudinal associations between symptoms in a controlled trial. J Subst Abuse Treat. 2012 Oct;43(3):291-302. doi: 10.1016/j.jsat.2011.12.010. Epub 2012 Mar 8. PMID 22406052
- [Result] Worley MJ, Trim RS, Tate SR, Hall JE, Brown SA. Service utilization during and after outpatient treatment for comorbid substance use disorder and depression. J Subst Abuse Treat. 2010 Sep;39(2):124-31. doi: 10.1016/j.jsat.2010.05.009. Epub 2010 Jul 3. PMID 20598832
- [Result] Mrnak-Meyer J, Tate SR, Tripp JC, Worley MJ, Jajodia A, McQuaid JR. Predictors of suicide-related hospitalization among U.S. veterans receiving treatment for comorbid depression and substance dependence: who is the riskiest of the risky? Suicide Life Threat Behav. 2011 Oct;41(5):532-42. doi: 10.1111/j.1943-278X.2011.00051.x. Epub 2011 Aug 4. PMID 21815915
- [Result] Worley MJ, Tate SR, Brown SA. Mediational relations between 12-Step attendance, depression and substance use in patients with comorbid substance dependence and major depression. Addiction. 2012 Nov;107(11):1974-83. doi: 10.1111/j.1360-0443.2012.03943.x. Epub 2012 Aug 10. PMID 22578037
- [Result] Worley MJ, Tate SR, McQuaid JR, Granholm EL, Brown SA. 12-step affiliation and attendance following treatment for comorbid substance dependence and depression: a latent growth curve mediation model. Subst Abus. 2013;34(1):43-50. doi: 10.1080/08897077.2012.691451. PMID 23327503
- [Result] Tripp JC, Skidmore JR, Cui R, Tate SR. Impact of Physical Health on Treatment for Co-occurring Depression and Substance Dependence. J Dual Diagn. 2013;9(3):10.1080/15504263.2013.806111. doi: 10.1080/15504263.2013.806111. PMID 24223036
- [Derived] Worley MJ, Tate SR, Granholm E, Brown SA. Mediated and moderated effects of neurocognitive impairment on outcomes of treatment for substance dependence and major depression. J Consult Clin Psychol. 2014 Jun;82(3):418-28. doi: 10.1037/a0036033. Epub 2014 Mar 3. PMID 24588403